CLINICAL TRIAL: NCT05334810
Title: A Multi-center, Open-lable, Single-arm Phase II Study to Evaluate the Efficacy and Safety of DP303c in Patients With HER2-positive Unresectable Locally Advanced, Relapsed, or Metastatic Breast Cancer
Brief Title: DP303c in Patients With HER2-positive Unresectable Locally Advanced, Relapsed, or Metastaticbreast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSA1501-CSP-005
Record Dates: First submitted 2022-03-27; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: HER2-positive Breast Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DP303c (Experimental): Eligible patients will be treated with DP303c at 3.0 mg/kg every 3 weeks.
  Interventions: Drug: DP303c

INTERVENTIONS:
Drug: DP303c — DP303c injection, 3.0 mg/kg, every 3 weeks.
  Other Names: DP303c treatment

SUMMARY:
This is a study of DP303c in patients with HER2-positive advanced breast cancer.

DETAILED DESCRIPTION:
This is a multi-center, open-lable, single-arm Phase II study to evaluate the efficacy and safety of DP303c in patients with HER2-positive unresectable locally advanced, relapsed, or metastatic breast cancer. Patients will be treated with DP303c injection at 3.0 mg/kg every 3 weeks. Patients will receive DP303c until disease progression, intolerable toxicity, withdrawal of informed consent, death, or any other reasons for treatment discontinuation, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary agreement to provide written informed consent;
2. Aged 18 to 75 years, male or female;
3. Patients with unresectable locally advanced, relapsed, or metastatic breast cancer confirmed by histology or cytology;
4. Received at least 2 lines of systemic anti-HER2 therapy for unresectable locally advanced, recurrent, or metastatic disease, and one of which is a trastuzumab-containing regimen, progression during or within 12 months of the end of prior (neo)adjuvant anti-HER2 therapy is considered one line of therapy.
5. Radiographic evidence of disease progression confirmed by the investigator during or after the most recent systemic treatment;
6. Sufficient tumor samples within 3 years are available for central lab to confirm the HER2 status;
7. Confirmed to be HER2 positive by central lab (HER2-positive is defined as IHC 3+ or IHC 2+ with ISH positive);
8. At least one measurable target lesion at the baseline according to the RECIST v1.1;
9. The Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
10. Left ventricular ejection fraction (LVEF) ≥50% of normal in echocardiogram (ECHO) or multi-gate detection scan (MUGA) within 4 weeks before the first administration of study drug;
11. The function of major organs must meet the following criteria within 7 days before enrollment (have not received blood transfusion, G-CSF, other hematopoietic stimulating factors or medical supportive treatments within 14 days before the first dose of study drug): absolute neutrophil count (ANC) ≥1.5×10^9 /L; platelet (PLT) ≥100×10^9 /L; hemoglobin ≥90 g/L; international normalized ratio (INR) or prothrombin time (PT) ≤1.5×the upper limit of normal (ULN) (not receiving anticoagulation), or patients receiving anticoagulation need to be within treatment target range and at a stable dose; activated partial thromboplastin time (APTT) ≤1.5×ULN; creatinine clearance rate>60 mL/min (calculated by Cockcroft-Gualt formula); total bilirubin ≤1.5×ULN, or ≤3×ULN for patients with Gilbert's syndrome; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN, or ≤5×ULN for patient with liver metastasis;
12. Life expectancy ≥ 3 months;
13. Women of childbearing age must have a negative pregnancy test prior to study entry;
14. Female and male patient of childbearing age must agree to take adequate contraceptive measures during the entire study period and through at least 6 months after the last dose of study drug.

Exclusion Criteria:

1. Pregnant or breastfeeding women；
2. History of DP303c treatment;
3. History of any other malignant tumors within five years (except for skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, cervical cancer in situ and other in situ tumors that have received radical resection and have not recurred);
4. Has not recovered from adverse reactions caused by previous anti-tumor treatments to ≤ grade 1 or baseline (refer to NCI CTCAE 5.0) (except for adverse reaction such as alopecia, pigmentation disorder and others which have no safety risk evaluated by the investigator);
5. Patients have received other clinical trial drugs within 4 weeks before the first dose of study drug (for small molecule targeted drugs, this time interval is required to be 2 weeks or 5 half-lives, whichever is longer);
6. Cytotoxic chemotherapy, radiotherapy and immunotherapy and other anti-tumor treatments within 4 weeks before the first dose of study drug; endocrine therapy and Chinese medicine treatments with anti-tumor indications within 2 weeks; or oral fluorouracil and small molecule targeted drugs within 2 weeks or 5 half-lives, whichever is longer;
7. Radical radiation therapy within 4 weeks before the first dose of study drug or palliative radiation therapy within 2 weeks before the first dose of study drug;
8. Underwent major surgery within 4 weeks and did not fully recover before the first dose of study drug;
9. The cumulative amount of previous exposure to anthracyclines has reached the following dosage: doxorubicin or liposomal doxorubicin >360 mg/m^2; epirubicin >720 mg/m^2; mitoxantrone>120 mg/m^2; idarubicin >90 mg/m^2; or other anthracyclines > 360 mg/m^2 of doxorubicin equivalent;
10. Untreated (including baseline findings) or unstable cerebral parenchymal metastasis, spinal cord metastasis or compression, and cancerous meningitis.
11. History of LVEF < 40%, symptomatic congestive heart failure (CHF), or associated toxicity leading to permanent discontinuation during previous treatments of trastuzumab or a drug containing a trastuzumab-like structure.
12. Serious or uncontrolled cardiovascular disease;
13. Serious or uncontrolled lung disease;
14. Symptomatic ascites or pleural effusion; patients who are clinically stable for at least 1 week after local treatment (including therapeutic pleural or abdominal puncture) are admitted;
15. Patients who currently have corneal diseases that require medication or surgical intervention, or have a history of serious corneal diseases, or are unwilling to stop wearing contact lenses during the study;
16. Peripheral neuropathy ≥ grade 2 (refer to NCI CTCAE 5.0) or history of ≥ grade 3 neurotoxicity (refer to NCI CTCAE 5.0);
17. Uncontrollable electrolyte imbalances include hypokalemia, hypocalcemia or hypomagnesemia (refer to NCI CTCAE 5.0, ≥2 grade);
18. Active infections requiring intravenous antibiotics, antivirals, or antifungals within 2 weeks before the first dose of study drug;
19. Active hepatitis B or C (HBsAg positive with HBV DNA >ULN, but patients with HBV DNA titer < 500 IU/mL after anti-HBV treatment could be enrolled; HCVAb positive with HCV RNA> ULN).
20. History of immunodeficiency diseases, including human immunodeficiency virus (HIV) positive;
21. Conditions requiring treatments with systemic corticosteroids or other immunosuppressive drugs within 2 weeks before the first dose of study drug, except for topical, ocular, intra-articular, intranasal, or inhaled corticosteroid therapy;
22. History of allergy to any components of study drug;
23. History of serious hypersensitivity to other monoclonal antibodies;
24. Suffering from a known mental illness, severe mental illness or poor compliance;
25. Treated with strong CYP3A inhibitors or strong CYP3A inducers within 14 days before the first dose of study drug;
26. Any disorders, treatments, or abnormalities in laboratory tests that may affect the overall treatments of patients in the study, increase the risk of patients, or interfere with the study results; or the investigator believes that participation in the study is not in the patient's best interest.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Baseline and every 6 weeks
  ORR is assessed by the Independent Review Committee (IRC) according to the Regulated Efficacy Criteria for Solid Tumors (RECIST) V1.1

SECONDARY OUTCOMES:
DOR | Baseline and every 6 weeks
  Duration of Response
PFS | Baseline and every 6 weeks
  Progression Free Survival

IPD SHARING:
Plan to Share IPD: No
Undecided.